CLINICAL TRIAL: NCT03835507
Title: Randomized, Double-blind, Safety and Efficacy of Recombinant Human Erythropoietin in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Seung Hyun Kim, MD, PhD, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HYNR-EPO
Record Dates: First submitted 2018-08-08; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Placebo Comparator): Inject Normal saline 100ml * 12 times (1month apart)
  Interventions: Drug: recombinant human erythropoietin(rhEPO)
- Low dose group (Experimental): Inject 500IU/kg of EPO mixed with normal saline 100ml * 12 times (1month apart)
  Interventions: Drug: recombinant human erythropoietin(rhEPO)
- High dose group (Experimental): Inject 750IU/kg of EPO mixed with normal saline 100ml * 12 times (1month apart)
  Interventions: Drug: recombinant human erythropoietin(rhEPO)

INTERVENTIONS:
Drug: recombinant human erythropoietin(rhEPO) — Injection of erythropoietin every months (total 12 months)

SUMMARY:
Erythropoietin is neuroprotective in animal models of neurodegenerative diseases including amyotrophic lateral sclerosis (ALS). The aim of this study was to determine the safety and feasibility of repetitive high-dose recombinant human erythropoietin (rhEPO) therapy in ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 to 80
* upper motor neuron signs and lower motor neuron signs were identified in neurological examination.
* Meet the revised El Escorial Criteria for clinically possible, probable-laboratory -supported, probable, definite ALS.
* Disease duration < 3 years (Within 3 years from symptom onset)
* ALSFRS-R score between 21 to 46
* Patient who can visit an outpatient under the aid of his or her own walking or caregivers.
* The person who have agreed in writing to participate in this clinical trial by themselves and the legal representative
* FVC over 50% at screening

Exclusion Criteria:

* Person who were not compatible with ALS
* Patient with PLS or PMA
* A group of patients who are concerned about the adverse effects of the drug administration (e.g. malignant hypertension,...)
* ALSFRS-R score below 20 at screening
* Ventilator user or Tracheostomy state patients at screening
* Gastrostomy state at screening
* FVC below 50% at screening or patient who cannot perform FVC test.
* EKG abnormality, history of coronary stent , CABG at screening
* Person who was given another clinical trial drug three months prior to screening.
* History of seizure/ epilepsy
* Abnormal renal function (serem creatinine > 2.0mg/dl)
* Abnormal liver function(AST/ALT/bilirubin over 2 times the upper normal limit
* Pregnant
* Bleeding tendency at screening
* Infectious disease at screening
* Drug sensitivity
* Person who injected erythropoietin 6 months prior to screening
* Malignant tumor
* Other neurological disease (stroke, parkinson's disease, dementia...)
* Psychological disease
* Hb more than 16g/dL

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-06-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
changes of ALSFRS-R score | Last visit [15th visit (15 months)]
  changes between score of ALSFRS-R at initial and study end point

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim HY, Moon C, Kim KS, Oh KW, Oh SI, Kim J, Kim SH. Recombinant human erythropoietin in amyotrophic lateral sclerosis: a pilot study of safety and feasibility. J Clin Neurol. 2014 Oct;10(4):342-7. doi: 10.3988/jcn.2014.10.4.342. Epub 2014 Oct 6. PMID 25324884
- [Result] Noh MY, Cho KA, Kim H, Kim SM, Kim SH. Erythropoietin modulates the immune-inflammatory response of a SOD1(G93A) transgenic mouse model of amyotrophic lateral sclerosis (ALS). Neurosci Lett. 2014 Jun 27;574:53-8. doi: 10.1016/j.neulet.2014.05.001. Epub 2014 May 10. PMID 24820540